CLINICAL TRIAL: NCT02663895
Title: A Pilot Study to Evaluate the Safety and Efficacy of Oral Treprostinil in the Treatment of Calcinosis in Patients With Systemic Sclerosis
Brief Title: Safety and Efficacy of Oral Treprostinil in the Treatment of Calcinosis in Patients With Systemic Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: United Therapeutics (Industry)
Responsible Party: Principal Investigator, Lorinda S Chung, Associate professor of medicine (Immunology & Rheumatology), Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 36140
Record Dates: First submitted 2016-01-19; First posted 2016-01-26 (Estimated); Results first posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Systemic Sclerosis; Calcinosis
MeSH Terms: conditions — Scleroderma, Systemic; Calcinosis | interventions — treprostinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Oral treprostinil (Experimental): Treprostinil 0.125 mg TID orally, which will be increased by 0.125 mg TID every 3 to 4 days as tolerated for 12 months
  Interventions: Drug: Oral treprostinil

INTERVENTIONS:
Drug: Oral treprostinil — Treprostinil 0.125 mg TID orally, which will be increased by 0.125 mg TID every 3 to 4 days as tolerated
  Other Names: Orenitram

SUMMARY:
This is a prospective open-label trial that will enroll 12 patients with systemic sclerosis (SSc) and at least one calcinotic lesion of the hands that is palpable on physical examination and also measureable on hand radiographs, at one single center. Each subject will receive treprostinil orally for 12 months, and follow-up evaluations will be performed every 3 months. Our main objective is to determine whether oral treprostinil is safe, and effective in reducing calcinosis in patients with SSc. We hypothesize that calcinosis is a result of microvascular injury and ischemic damage, and that therefore treprostinil may be beneficial in the treatment of calcinosis in patients with SSc.

DETAILED DESCRIPTION:
1. Background:

   Calcinosis cutis is the deposition of calcium in the skin and subcutaneous tissues. It is a common and potentially debilitating manifestation of systemic sclerosis (SSc), affecting almost one quarter of these patients. Several studies have found an association between calcinosis and vascular manifestations of SSc including digital ulcers (DU), and acro-osteolysis. The investigators confirmed this in a retrospective multi-center international cohort study of 5280 patients with SSc where DUs were the strongest predictor of calcinosis in multivariate analysis (OR 3.7, 95%CI 2.6-5.3, p<0.0001).

   Treprostinil delivered by continuous subcutaneous infusion was effective in both the healing and prevention of DU in patients with SSc in an open-label, single-center clinical trial of 5 (of 12) patients who were able to tolerate the medication. A study of 148 subjects with DU showed that the administration of oral treprostinil up to 16 mg twice daily for 20 weeks was associated with a small but statistically insignificant reduction in net ulcer burden in comparison to placebo. Additionally, preliminary observations in the Pulmonary Hypertension Assessment and Recognition of Outcomes in Scleroderma (PHAROS) registry have found that two patients with SSc-PAH and calcinosis treated with subcutaneous treprostinil for PAH experienced approximately 50% radiographic improvement in their calcinosis lesions after 6 months of therapy.

   The investigators developed and validated a novel radiographic scoring system to assess the severity of calcinosis affecting the hands of patients with SSc that accounts for area coverage, density, and anatomic location. This scoring system is feasible and was found to have excellent intra- and inter-rater reliability with intra-class correlation coefficients (ICC) of .93 (.89-.97) and .89 (.86-.92), respectively.

   Given that calcinosis is a frequent, debilitating complication of SSc associated with digital vascular ischemia with no effective therapies, a clinical trial, using novel outcome measures, testing the safety and efficacy of a powerful vasodilator for the treatment of calcinosis is warranted.
2. Primary/Secondary objectives:

   Our main objective is to conduct an open-label proof-of-concept study with the primary and secondary endpoints entered elsewhere.
3. Hypothesis:

   The investigators hypothesize that calcinosis is a result of microvascular injury and ischemic damage, and that therefore treprostinil may be beneficial in the treatment of calcinosis in patients with SSc.
4. Study design:

   This prospective open-label trial will enroll 12 patients with SSc and at least one calcinotic lesion of the hands that is palpable on physical examination and also measureable on hand radiographs. Each subject will undergo a screening evaluation 4 weeks before treatment with the study drug is initiated. Each subject will receive treprostinil 0.125 mg TID orally, which will be increased by 0.125 mg TID every 3 to 4 days as tolerated. Follow-up evaluations will be performed every 3 months over a 12-month period of time.
5. Study population:

   The population for this study will consist of adult SSc patients with evidence of at least one calcinotic lesion of the hands that is palpable on physical examination and also measureable on hand radiographs. Inclusion and exclusion criteria have been entered elsewhere.
6. Description of the treatment:

   United Therapeutics will provide treprostinil labeled for investigational use. The Sponsor/Investigator of the trial will ensure maintenance of complete and accurate records of the receipt, dispensation, and disposal or return of all trial drug in accordance with Title 21 Code of Federal Regulations (C.F.R.), Part 312.57 and 312.62 and United Therapeutics requirements.

   Treprostinil Treprostinil (Orenitram) is a prostacyclin vasodilator indicated for the treatment of pulmonary arterial hypertension (WHO Group 1) to improve exercise capacity. The molecular formula is C23H34O5C4H11NO2, and its molecular weight is 495.65. Orenitram is an extended release osmotic tablet for oral administration, and it is formulated as the diolamine salt of treprostinil, a tricyclic benzindene analogue of prostacyclin. It is available in the following four strengths: 0.125 mg (white tablet imprinted with UT 0.125), 0.25 mg (green tablet imprinted with UT 0.25), 1 mg (yellow tablet imprinted with UT 1), and 2.5 mg (pink tablet imprinted with UT 2.5). The formulations also contain xylitol, maltodextrin, sodium lauryl sulfate, magnesium stearate, cellulose acetate, triethyl citrate, polyvinyl alcohol, titanium dioxide, polyethylene glycol, and talc. In addition tablets may contain colorants FD&C Blue 2, iron oxide yellow, and iron oxide red. The imprinting ink contains shellac glaze, ethanol, isopropyl alcohol USP, iron oxide black, n-butyl alcohol, propylene glycol, and ammonium hydroxide.

   Mechanism of Action The major pharmacologic actions of treprostinil are direct vasodilation of pulmonary and systemic arterial vascular beds, inhibition of platelet aggregation, and inhibition of smooth muscle cell proliferation.

   Storage Treprostinil must be stored at 25°C (77°F); excursions 15°C to 30°C (59°F to 86°F). For further details, see the Investigator Brochure and the Orenitram Package Insert.

   Dosage and Administration Initiate treprostinil at 0.125 mg TID (every 8 ± 2 h), with dose escalation of an additional 0.125 mg TID every 3 to 4 days as tolerated. No dose changes will be allowed for 5 days before the month 12 visit. Give with food, swallow tablets whole, and use only intact tablets; do not crush, split, or chew. The maximum dose, dose escalation or titration will be done at the Investigator's discretion based upon individual subject tolerability. Patients with mild hepatic impairment (Child Pugh Class A) should initiate treprostinil at 0.125 mg TID, and increment at 0.125 mg TID every 6 to 8 days.[8]

   Criteria for Treatment Discontinuation

   Treatment will be discontinued in the following circumstances:
   * Patients who wish to withdraw from further participation
   * Patients with a serious or life-threatening adverse event that in the opinion of the investigator is directly attributable to the study drug
   * The patient deviated from the protocol
   * The patient's behavior is likely to undermine the validity of his / her results
   * Patients who have a positive pregnancy test during the study
   * Patients who develop any condition that in the opinion of the investigator could be worsened by further treatment with the study drug

   Criteria for Stopping Rules The study may be stopped at any time if, in the opinion of the Investigator and / or Sponsor, continuation of the study represents a serious medical risk to the subjects. This may include, but is not limited to, the presence of serious, life-threatening, or fatal adverse events or adverse events that are unacceptable in nature, severity, or frequency. The Sponsor reserves the right to discontinue the study for any reason at any time.
7. Estimated duration: 12 months
8. Time and events schedule and description of assessments:

   What will happen at each visit?

   Screening Visit (1 month prior to treatment):
   * Informed consent
   * Review of inclusion and exclusion criteria
   * Complete medical history including scleroderma diagnosis
   * Review of concomitant medications
   * Complete physical examination including examination of calcinosis, digital ulcers, vital signs, height/weight, and Modified Rodnan skin score (MRSS)
   * Electrocardiogram (EKG)
   * Laboratory tests: CBC with differential, comprehensive metabolic panel, and urinalysis
   * Urine pregnancy test (females of child bearing potential only)
   * Review of adverse events

   Baseline Visit (0 month):
   * Review of concomitant medications
   * Complete physical examination with vital signs, and MRSS
   * Examination of calcinosis and digital ulcers
   * Laboratory tests: CBC with differential, comprehensive metabolic panel, and urinalysis
   * Urine pregnancy test (females of child bearing potential only)
   * Questionnaires: SHAQ, Cochin hand functional scale, SF-36 assessment of health status, Mawdsley Calcinosis Questionnaire, Physician/Patient Global Assessment of calcinosis severity, and Raynaud's Condition Score.
   * Review of adverse events
   * Study drug dispense/return
   * Radiological assessment of calcinosis
   * Skin biopsy
   * Blood for biomarker analyses
   * SPY assessment of superficial blood flow
   * XtremeCT II scan

   At 3 months visit:
   * Review of concomitant medications
   * Examination of calcinosis and digital ulcers
   * Urine pregnancy test (females of child bearing potential only)
   * Questionnaires: SHAQ, Cochin hand functional scale, SF-36 assessment of health status, Mawdsley Calcinosis Questionnaire, Physician/Patient Global Assessment of calcinosis severity, and Raynaud's Condition Score.
   * Blood for biomarker analyses
   * Review of adverse events
   * Study drug dispense/return

   At 6 months visit:
   * Review of concomitant medications
   * Examination of calcinosis and digital ulcers
   * Complete physical examination with vital signs, and MRSS
   * Laboratory tests: CBC with differential, comprehensive metabolic panel, and urinalysis
   * Urine pregnancy test (females of child bearing potential only)
   * Questionnaires: SHAQ, Cochin hand functional scale, SF-36 assessment of health status, Mawdsley Calcinosis Questionnaire, Physician/Patient Global Assessment of calcinosis severity, and Raynaud's Condition Score.
   * Review of adverse events
   * Study drug dispense/return

   At 9 months visit:
   * Review of concomitant medications
   * Examination of calcinosis and digital ulcers
   * Urine pregnancy test (females of child bearing potential only)
   * Questionnaires: SHAQ, Cochin hand functional scale, SF-36 assessment of health status, Mawdsley Calcinosis Questionnaire, Physician/Patient Global Assessment of calcinosis severity, and Raynaud's Condition Score.
   * Review of adverse events
   * Study drug dispense/return

   At 12 months visit:
   * Review of concomitant medications
   * Examination of calcinosis and digital ulcers
   * Urine pregnancy test (females of child bearing potential only)
   * Questionnaires: SHAQ, Cochin hand functional scale, SF-36 assessment of health status, Mawdsley Calcinosis Questionnaire, Physician/Patient Global Assessment of calcinosis severity, and Raynaud's Condition Score.
   * Review of adverse events
   * Study drug dispense/return
   * Complete physical examination with vital signs, and MRSS
   * Laboratory tests: CBC with differential, comprehensive metabolic panel, and urinalysis
   * Radiological assessment of calcinosis
   * Skin biopsy
   * Blood for biomarker analyses
   * SPY assessment of superficial blood flow
   * EKG

   Description of assessments:

   Medical history including SSc: Significant past or present illnesses, current prescription or nonprescription medications (including vitamins and herbal products), and history of allergies or idiosyncratic responses to drugs should be noted.

   Physical examination: A complete physical examination will be conducted by a physician at Screening, 6 months, and at end of study. Any significant changes to the subject's medical condition, physical examination, and concomitant medications should be documented throughout the course of the study. Any untoward medical experience should be recorded as an adverse event.

   Examination of calcinosis and digital ulcers: Investigator will perform a thorough clinical examination looking for calcinotic deposits at each visit. The investigators will use case report forms with picture images of the hands to record calcinosis and digital ulcers at each evaluation. The investigators will define digital ulcer as an area with visually discernable depth and a loss of continuity of epithelial coverage in the volar aspect of the finger and distal from the proximal interphalangeal joints, which could be denuded (active) or covered by a scab or necrotic tissue (indeterminate). At each visit, the status of each digital ulcer will be rated as "A," a current active digital ulcer, "H", a completely healed ulcer, or "I," an ulcer with indeterminate status, as previously defined.

   Vital Signs: Systolic and diastolic blood pressure, heart rate, respiratory rate, and temperature (°C) will be measured prior to assessments and after sitting for 5 minutes at screening, baseline, 6 months, and 12 months. Vital signs should also be assessed in the case of abnormal clinical signs and symptoms.

   Electrocardiogram (ECG): Twelve-lead ECGs will be recorded after at least 5 minutes rest in the semi-recumbent position at screening and at the end of the study at 12 months. Recordings should include lead II as a rhythm strip and contain at least 5 QRS complexes. ECG parameters collected (after at least 5 minutes rest) include heart rate, and PR interval, QT interval, QRS duration and any clinically significant abnormalities.

   Laboratory tests: Blood and urine samples for the measurement and evaluation of CBC, CMP, and urinalysis (UA) will be collected at screening, 6 months and at the end of the study, and analyzed at Stanford laboratory.

   Urine pregnancy test: urine beta-HCG will be measured in all female in reproductive age at all visits.

   Radiological examination of calcinosis: Patients will have plain radiographs of the hands at baseline and at 1 year.

   Scleroderma Health Assessment Questionnaire (SHAQ): The SHAQ is a patient self-administered instrument, which has been previously validated in SSc and demonstrates meaningful clinical changes in the course of the disease over time. It is comprised of the HAQ-DI, a self-administered 20-question instrument that assesses a patient's level of functional ability and five scleroderma visual analogue scale (VAS) measurements to evaluate symptoms specific to SSc.

   Cochin Hand Function Scale (CHFS): CHFS is a questionnaire derived from 18 validated questions to assess functional disability and handicap due to hand involvement in rheumatoid arthritis. Each answer is scored on a scale of 0 (no difficulty) to 5 (impossible to do), with a maximum score of 90. A higher score indicates worse disability or handicap. The CHFS has been demonstrated as a reliable and valid assessment of hand function at the activity level in persons with SSc.

   Mawdsley Calcinosis Questionnaire: The content of this questionnaire is patient-generated and includes 17 questions related to the impact of calcinosis rated from 0 (no limitation) to 10 (worst limitation possible).

   The Medical Outcomes Study 36-Item Short Form Health Survey (SF-36): The SF-36 is one of the most widely used instruments to assess quality of life in patients with systemic illnesses. It is a self-administered questionnaire covering eight areas: physical function, physical role, bodily pain, general health, vitality, social function, emotional role, and mental health. For each area, the score ranges from 0 (poorer health status) to 100 (better health status).

   Patient and Physician global assessments: Patients and physicians will each independently rate the severity of calcinosis on a 10 cm VAS. The term "severity" will be used to measure the extent of disease activity and associated disability or discomfort the patient experiences during the indicated time period.

   Raynaud's Condition Score (RCS): The investigators will measure changes in Raynaud's phenomenon (RP) by using the RCS, a self-assessment of RP activity using a 0-10 ordinal scale. The RCS incorporates the cumulative daily frequency, duration, severity, and impact of RP attacks.

   Modified Rodnan Skin Score (mRSS): The mRSS measures skin tightness and is the sum of scores from 17 surface anatomic areas (fingers, hands, forearms, arms, feet, legs, and thighs bilaterally, and face, chest, and abdomen singly) rated on a 0-3 scale (0=normal skin; 1=mild thickness; 2=moderate thickness; 3=severe thickness with inability to pinch the skin into a fold). The skin score will be the sum of the individual skin assessment scores and ranges from 0 (best possible outcome) to 51 (worst possible outcome).

   Skin biopsies: The investigators will collect two side-by-side skin samples to assess for vascular changes on histopathology and gene expression changes following treatment with treprostinil: one at baseline and one at the end of the study. This part of the study will be optional for participating patients. Skin biopsies will be obtained from a standard site on the forearm (extensor surface of forearm approximately 10 cm proximal to the olecranon, which is chosen for its uniform involvement in patients with SSc). Two adjacent 5 mm punch biopsies (taken full thickness to subcutaneous fat) will be harvested from the site. This involves selecting an area to biopsy and wiping the skin with alcohol. Next, 1-2 cc of lidocaine with 1:100,000 epinephrine is introduced into the skin using a 30G needle. Two punch biopsies will then be taken and processed as described in appendix I. Next, the wound will be sutured with 1-2 4.0 nylon sutures. Wounds will be dressed with polysporin and a bandage. Verbal wound care instructions will be given. The first biopsy will be bisected: one half will be flash frozen in liquid nitrogen and half will be embedded in paraffin. The second biopsy will also be bisected: one half will be placed in RNA later, and the other half will be placed in a cryo-tube.

   Research blood: The investigators will collect serum and peripheral blood samples to assess changes in vascular and SSc-associated biomarkers following treatment with treprostinil. Blood samples for the assessment of biomarkers will be drawn at baseline, 3 months, and end of study visit. Please see appendix for a complete list of biomarkers.

   SPY: The SPY Near-Infrared Perfusion Assessment System (distributed by LifeCell Corp., Branchburg, N.J.; manufactured by Novadaq Technologies Inc., Richmond, BC, Canada) is an imaging technology that utilizes indocyanine green (ICG), and allows real-time visual assessment of superficial blood flow.

   XtremeCT II scan: The latest-generation high-resolution peripheral quantitative computed tomography (HR-pQCT) XtremeCT II scan is a novel technology with dramatically improved spatial resolution. It is able to define the cortical and trabecular surfaces of the bones in a three-dimensional fashion, and therefore provides information on bone microarchitecture as well as bone density. The XtremeCT II machine at Stanford University is one of 10 in the United States.

   Safety: During the study, the primary assessment of safety will be changes in vital signs, clinical laboratory parameters, EKG, and the development of adverse events.
9. Safety monitoring and reporting

   Definitions:

   Adverse Event (AE): An AE is any untoward medical experience occurring to a subject during a clinical trial whether or not it is related to the study drug. An AE may include an intercurrent illness, injury, or any other concomitant impairment of the subject's health, as well as abnormal laboratory findings if deemed to have clinical significance. AEs may also include worsening of an existing symptom or condition or post-treatment events that occur as a result of protocol-mandated procedures.

   Severe Adverse Event (SAE): A SAE is an AE occurring at any dose that results in any of the following outcomes:
   * Death
   * A life-threatening AE
   * Inpatient hospitalization or prolongation of existing hospitalization
   * A persistent or significant disability / incapacity
   * A congenital anomaly / birth defect

   In addition, important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the subject and require medical / surgical intervention to prevent one of the outcomes listed above. Examples of such medical events include allergic bronchospasm requiring intensive treatment in an emergency room or at home, blood dyscrasias or convulsions that do not result in hospitalization, or the development of drug dependency or drug abuse. Life threatening means that the subject was, in the view of the Investigator, at immediate risk of death from the event as it occurred. It does not mean that the event, had it occurred in a more severe form, might have caused death.

   Reporting Responsibilities:

   In the event of an adverse event, the first concern will be for the safety of the patients.

   Investigators are required to collect and document all adverse events (AEs) and non-related serious adverse events (SAEs). All SAEs, regardless of expectedness or causality, must be reported to the Sponsor by fax (+ 1 919-313-1297 or other appropriate number) within 24 hours of awareness. A completed SAE report form along with any relevant hospital records and autopsy reports should be faxed to the Drug Safety Department at United Therapeutics Corporation. A follow-up SAE report form must be forwarded to the Drug Safety Department at United Therapeutics Corporation within 48 hours of the receipt of any new / updated information. The Investigator must also promptly notify their Investigational Review Board (IRB) or Ethics Committee (EC) of the SAE, including any follow-up information, in accordance with applicable national regulations and guidelines set forth by the IRB or EC. All documents related to AEs (serious, non serious, related, or not) will be readily available for review, should the need arise.

   An AE or SAE occurring during the study must be documented in the subject's source documents and on the appropriate CRF page. Information relating to the AE such as onset and cessation date and times, intensity, seriousness, relationship to study drug, and outcome is also to be documented in the CRF. Where possible, AEs should be recorded using standard medical terminology. If several signs or symptoms are clearly related to a medically defined diagnosis or syndrome, the diagnosis or syndrome should be recorded on the CRF page, not the individual signs and symptoms.

   All AEs should be followed until either resolution (or return to normal or baseline values), until they are judged by the Investigator to no longer be clinically significant, or for at least 4 weeks if the AE extends beyond the final visit. All SAEs that occur during the study will be followed until resolution, death, or the subject is lost to follow-up even if they are ongoing more than 4 weeks after completion of the final visit. Supplemental measurements and / or evaluations may be necessary to investigate fully the nature and / or causality of an AE or SAE. This may include additional laboratory tests, diagnostic procedures, or consultation with other healthcare professionals. CRF pages should be updated.
10. Statistical Considerations

Statistical analysis:

Descriptive statistics and frequency distributions of all variables of interest will be reported as proportions (%) for categorical variables and as mean ± standard deviation or median (range) for continuous variables. Baseline to 12 month differences and 95% confidence intervals will be calculated for scored outcomes (x-ray score, MRSS, physician's global assessment by VAS, and quality of life measurements). For the primary efficacy endpoint, mean change and standard deviation in calcinosis burden assessed by radiograph from baseline to 12-month visit, the investigators will use Student's t-test. The mean rate of change of calcinosis in radiograph will be calculated with the following formula: (Year 1 XR score - Baseline XR score)/time. XR score is defined as: sum of scores for 22 weighted areas affecting each hand: %area coverage (0-100) X density (1-3) X weight for each area.

Sample size calculation:

The investigators will need 9 paired radiographs (9 patients) at 1-year to provide >80% power to detect a mean change in x-ray score of 12.0 (equivalent to a minimally significant change in score of 25%) with a SD of 8.2 with moderate correlation r=0.5 using a two-sided test at alpha 0.05 level. The investigators estimate a 15% dropout rate based on prior clinical trials. Hence, the total number of subjects needed to obtain 9/0.85 subjects who complete the study is 11 subjects. Also, due to the small sample size, the investigators plan to use Wilcoxon signed rank test to analyze the effects. Thus, the investigators anticipate losing about 10% of power due to using a non-parametric test. As a result, the sample size is further adjusted to 11/0.9 = 12. Statistical significance will be defined as p ≤ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Age > 18 years of age
* Diagnosis of limited or diffuse cutaneous systemic sclerosis (SSc) according to the revised 2013 ACR/EULAR classification criteria for SSc
* Radiological and physical examination evidence of at least one subcutaneous calcium deposition in the hands that is clinically apparent as part of routine clinical care.
* If female of childbearing potential, the patient must have a negative pregnancy test at screening and baseline visits
* Oral corticosteroids (≤ 10 mg/day of prednisone or equivalent) and NSAIDs are permitted if the patient is on a stable dose regimen for ≥ 2 weeks prior to screening and throughout the study
* Calcium channel blockers, alpha-1-antagonists, ACE-inhibitors, angiotensin receptor blockers, and protein-pump inhibitors are permitted as long as the doses are stable for 4 weeks prior to screening and throughout the study
* Women of childbearing potential must agree to use adequate contraception when sexually active with any combination of at least 2 effective methods of birth control (except for women who have a partner who is sterile, i.e. due to vasectomy)

Exclusion Criteria:

* Rheumatic disease other than SSc
* Patients with pulmonary arterial hypertension (PAH), NYHA Class III or IV, as determined by right heart catheterization or on PAH approved medications for PAH
* Patients with moderate or severe hepatic impairment (Child Pugh Class C), or transaminase elevation (ALT or AST) > 3 x the upper limit of normal at screening visit
* Patients with diverticulosis
* Hemoglobin < 75% of the lower limit of the normal range
* Systolic blood pressure < 95 mmHg or diastolic blood pressure < 50 mmHg
* Patients who are hemodynamically unstable, or have acute renal, cardiac or pulmonary failure, or any life-threatening condition.
* Concurrent malignancy except non-melanoma skin cancers
* Patients receiving specific (sildenafil, tadalafil) or unspecific phosphodiesterase-5 inhibitors (dipyridamole, theophylline), endothelin receptor antagonists, prostanoids, riociguat, or NO donors (nitrates) within 4 weeks of screening
* Patients receiving bisphosphonates, warfarin, colchicine, minocycline, intravenous immunoglobulins, or biological agents including abatacept or rituximab within 4 weeks of screening
* Patients receiving local treatments for calcinosis including surgical removal or intralesional steroid injections within 12 weeks of screening or throughout the study.
* Patients who have participated in another clinical trial of an investigative agent within 30 days of screening (or 5 half-lives of the investigational drug, whichever is longer)
* Pregnant or nursing women
* Patients with a history of drug or alcohol abuse within 6 months of screening
* Any medical condition that, in the opinion of the investigator, might interfere with the subject's participation in the study or poses an added risk for the subject
* Inability to comply with study and follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2016-10; Primary Completion 2020-05-13 (Actual); Study Completion 2020-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lorinda S Chung, MD, MS, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Avouac J, Mogavero G, Guerini H, Drape JL, Mathieu A, Kahan A, Allanore Y. Predictive factors of hand radiographic lesions in systemic sclerosis: a prospective study. Ann Rheum Dis. 2011 Apr;70(4):630-3. doi: 10.1136/ard.2010.134304. Epub 2010 Dec 3. PMID 21131648
- [Background] Koutaissoff S, Vanthuyne M, Smith V, De Langhe E, Depresseux G, Westhovens R, De Keyser F, Malghem J, Houssiau FA. Hand radiological damage in systemic sclerosis: comparison with a control group and clinical and functional correlations. Semin Arthritis Rheum. 2011 Apr;40(5):455-60. doi: 10.1016/j.semarthrit.2010.06.008. Epub 2010 Sep 22. PMID 20864145
- [Background] Johnstone EM, Hutchinson CE, Vail A, Chevance A, Herrick AL. Acro-osteolysis in systemic sclerosis is associated with digital ischaemia and severe calcinosis. Rheumatology (Oxford). 2012 Dec;51(12):2234-8. doi: 10.1093/rheumatology/kes214. Epub 2012 Aug 25. PMID 22923763
- [Background] Chung L, Fiorentino D. A pilot trial of treprostinil for the treatment and prevention of digital ulcers in patients with systemic sclerosis. J Am Acad Dermatol. 2006 May;54(5):880-2. doi: 10.1016/j.jaad.2006.02.004. PMID 16635673
- [Background] Chung L, Valenzuela A, Fiorentino D, Stevens K, Li S, Harris J, Hutchinson C, Assassi S, Beretta L, Lakshminarayanan S, Rodriguez-Reyna TS, Denton CP, Taillefer RG, Herrick AL, Baron M; Scleroderma Clinical Trials Consortium Calcinosis Working Group. Validation of a novel radiographic scoring system for calcinosis affecting the hands of patients with systemic sclerosis. Arthritis Care Res (Hoboken). 2015 Mar;67(3):425-30. doi: 10.1002/acr.22434. PMID 25155948
- [Background] Tapson VF, Jing ZC, Xu KF, Pan L, Feldman J, Kiely DG, Kotlyar E, McSwain CS, Laliberte K, Arneson C, Rubin LJ; FREEDOM-C2 Study Team. Oral treprostinil for the treatment of pulmonary arterial hypertension in patients receiving background endothelin receptor antagonist and phosphodiesterase type 5 inhibitor therapy (the FREEDOM-C2 study): a randomized controlled trial. Chest. 2013 Sep;144(3):952-958. doi: 10.1378/chest.12-2875. PMID 23669822
- [Background] Baron M, Chung L, Gyger G, Hummers L, Khanna D, Mayes MD, Pope JE, Shah AA, Steen VD, Steele R, Tatibouet S, Herrick A, Muller-Ladner U, Hudson M. Consensus opinion of a North American Working Group regarding the classification of digital ulcers in systemic sclerosis. Clin Rheumatol. 2014 Feb;33(2):207-14. doi: 10.1007/s10067-013-2460-7. Epub 2013 Dec 20. PMID 24357325
- [Background] Fries JF, Spitz P, Kraines RG, Holman HR. Measurement of patient outcome in arthritis. Arthritis Rheum. 1980 Feb;23(2):137-45. doi: 10.1002/art.1780230202. PMID 7362664
- [Background] Poole JL, Williams CA, Bloch DA, Hollak B, Spitz P. Concurrent validity of the Health Assessment Questionnaire Disability Index in Scleroderma. Arthritis Care Res. 1995 Sep;8(3):189-93. doi: 10.1002/art.1790080312. PMID 7654804
- [Background] Steen VD, Medsger TA Jr. The value of the Health Assessment Questionnaire and special patient-generated scales to demonstrate change in systemic sclerosis patients over time. Arthritis Rheum. 1997 Nov;40(11):1984-91. doi: 10.1002/art.1780401110. PMID 9365087
- [Background] Duruoz MT, Poiraudeau S, Fermanian J, Menkes CJ, Amor B, Dougados M, Revel M. Development and validation of a rheumatoid hand functional disability scale that assesses functional handicap. J Rheumatol. 1996 Jul;23(7):1167-72. PMID 8823687
- [Background] Brower LM, Poole JL. Reliability and validity of the Duruoz Hand Index in persons with systemic sclerosis (scleroderma). Arthritis Rheum. 2004 Oct 15;51(5):805-9. doi: 10.1002/art.20701. PMID 15478150
- [Background] Danieli E, Airo P, Bettoni L, Cinquini M, Antonioli CM, Cavazzana I, Franceschini F, Cattaneo R. Health-related quality of life measured by the Short Form 36 (SF-36) in systemic sclerosis: correlations with indexes of disease activity and severity, disability, and depressive symptoms. Clin Rheumatol. 2005 Feb;24(1):48-54. doi: 10.1007/s10067-004-0970-z. Epub 2004 Aug 6. PMID 15300468
- [Background] Del Rosso A, Boldrini M, D'Agostino D, Placidi GP, Scarpato A, Pignone A, Generini S, Konttinen Y, Zoppi M, Vlak T, Placidi G, Matucci-Cerinic M. Health-related quality of life in systemic sclerosis as measured by the Short Form 36: relationship with clinical and biologic markers. Arthritis Rheum. 2004 Jun 15;51(3):475-81. doi: 10.1002/art.20389. PMID 15188336
- [Background] Khanna D, Furst DE, Wong WK, Tsevat J, Clements PJ, Park GS, Postlethwaite AE, Ahmed M, Ginsburg S, Hays RD; Scleroderma Collagen Type 1 Study Group. Reliability, validity, and minimally important differences of the SF-6D in systemic sclerosis. Qual Life Res. 2007 Aug;16(6):1083-92. doi: 10.1007/s11136-007-9207-3. Epub 2007 Apr 3. PMID 17404896
- [Background] Kosinski M, Keller SD, Hatoum HT, Kong SX, Ware JE Jr. The SF-36 Health Survey as a generic outcome measure in clinical trials of patients with osteoarthritis and rheumatoid arthritis: tests of data quality, scaling assumptions and score reliability. Med Care. 1999 May;37(5 Suppl):MS10-22. doi: 10.1097/00005650-199905001-00002. PMID 10335740
- [Background] Kosinski M, Keller SD, Ware JE Jr, Hatoum HT, Kong SX. The SF-36 Health Survey as a generic outcome measure in clinical trials of patients with osteoarthritis and rheumatoid arthritis: relative validity of scales in relation to clinical measures of arthritis severity. Med Care. 1999 May;37(5 Suppl):MS23-39. doi: 10.1097/00005650-199905001-00003. PMID 10335741
- [Background] Rannou F, Boutron I, Jardinaud-Lopez M, Meric G, Revel M, Fermanian J, Poiraudeau S. Should aggregate scores of the Medical Outcomes Study 36-item Short Form Health Survey be used to assess quality of life in knee and hip osteoarthritis? A national survey in primary care. Osteoarthritis Cartilage. 2007 Sep;15(9):1013-8. doi: 10.1016/j.joca.2007.02.012. Epub 2007 Mar 26. PMID 17387025
- [Background] Rannou F, Poiraudeau S, Berezne A, Baubet T, Le-Guern V, Cabane J, Guillevin L, Revel M, Fermanian J, Mouthon L. Assessing disability and quality of life in systemic sclerosis: construct validities of the Cochin Hand Function Scale, Health Assessment Questionnaire (HAQ), Systemic Sclerosis HAQ, and Medical Outcomes Study 36-Item Short Form Health Survey. Arthritis Rheum. 2007 Feb 15;57(1):94-102. doi: 10.1002/art.22468. PMID 17266096
- [Background] Strand V. Longer term benefits of treating rheumatoid arthritis: assessment of radiographic damage and physical function in clinical trials. Clin Exp Rheumatol. 2004 Sep-Oct;22(5 Suppl 35):S57-64. PMID 15552516
- [Background] Ware JE Jr, Sherbourne CD. The MOS 36-item short-form health survey (SF-36). I. Conceptual framework and item selection. Med Care. 1992 Jun;30(6):473-83. PMID 1593914
- [Background] Merkel PA, Herlyn K, Martin RW, Anderson JJ, Mayes MD, Bell P, Korn JH, Simms RW, Csuka ME, Medsger TA Jr, Rothfield NF, Ellman MH, Collier DH, Weinstein A, Furst DE, Jimenez SA, White B, Seibold JR, Wigley FM; Scleroderma Clinical Trials Consortium. Measuring disease activity and functional status in patients with scleroderma and Raynaud's phenomenon. Arthritis Rheum. 2002 Sep;46(9):2410-20. doi: 10.1002/art.10486. PMID 12355489
- [Background] Clements P, Lachenbruch P, Siebold J, White B, Weiner S, Martin R, Weinstein A, Weisman M, Mayes M, Collier D, et al. Inter and intraobserver variability of total skin thickness score (modified Rodnan TSS) in systemic sclerosis. J Rheumatol. 1995 Jul;22(7):1281-5. PMID 7562759
- [Background] Clements PJ, Lachenbruch PA, Seibold JR, Zee B, Steen VD, Brennan P, Silman AJ, Allegar N, Varga J, Massa M, et al. Skin thickness score in systemic sclerosis: an assessment of interobserver variability in 3 independent studies. J Rheumatol. 1993 Nov;20(11):1892-6. PMID 8308774
- [Background] Furst DE, Clements PJ, Steen VD, Medsger TA Jr, Masi AT, D'Angelo WA, Lachenbruch PA, Grau RG, Seibold JR. The modified Rodnan skin score is an accurate reflection of skin biopsy thickness in systemic sclerosis. J Rheumatol. 1998 Jan;25(1):84-8. PMID 9458208
- [Background] Brooks D. Perfusion Assessment with the SPY System after Arterial Venous Reversal for Upper Extremity Ischemia. Plast Reconstr Surg Glob Open. 2014 Aug 7;2(7):e185. doi: 10.1097/GOX.0000000000000138. eCollection 2014 Jul. PMID 25426368
- [Background] van den Hoogen F, Khanna D, Fransen J, Johnson SR, Baron M, Tyndall A, Matucci-Cerinic M, Naden RP, Medsger TA Jr, Carreira PE, Riemekasten G, Clements PJ, Denton CP, Distler O, Allanore Y, Furst DE, Gabrielli A, Mayes MD, van Laar JM, Seibold JR, Czirjak L, Steen VD, Inanc M, Kowal-Bielecka O, Muller-Ladner U, Valentini G, Veale DJ, Vonk MC, Walker UA, Chung L, Collier DH, Csuka ME, Fessler BJ, Guiducci S, Herrick A, Hsu VM, Jimenez S, Kahaleh B, Merkel PA, Sierakowski S, Silver RM, Simms RW, Varga J, Pope JE. 2013 classification criteria for systemic sclerosis: an American College of Rheumatology/European League against Rheumatism collaborative initiative. Arthritis Rheum. 2013 Nov;65(11):2737-47. doi: 10.1002/art.38098. Epub 2013 Oct 3. PMID 24122180
- [Derived] Chung MP, Valenzuela A, Li S, Catanese B, Stevens K, Fiorentino D, Strand V, Chung L. A pilot study to evaluate the safety and efficacy of treprostinil in the treatment of calcinosis in systemic sclerosis. Rheumatology (Oxford). 2022 May 30;61(6):2441-2449. doi: 10.1093/rheumatology/keab810. PMID 34718447

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral Treprostinil: Treprostinil 0.125 mg three times daily (TID), increased by 0.125 mg TID every 3 to 4 days as tolerated for 12-month period of time.
Period: Overall Study
Arm/Group | Oral Treprostinil
Started | 12
Completed | 5
Not Completed | 7
Not completed — Adverse Event | 3
Not completed — Physician Decision | 2
Not completed — Progressive Systemic Sclerosis (SSc) | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Oral Treprostinil
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 55 [35 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 9
  Hispanic | 2
  African-American | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12
Disease Duration from First non-Raynaud symptom [Median (Full Range); unit: years] | 12.3 [5.6 to 20.5]
Ever Smoker [Count of Participants; unit: Participants] | 4
Presence of diffuse cutaneous disease [Count of Participants; unit: Participants] | 6
Calcinosis in Radiograph [Median (Full Range); unit: score on a scale] — Assessed by the Scleroderma Clinical Trial Consortium (SCTC) radiographic scoring system. Historical average SCTC scores in this patient population have ranged from 4.08 to 472.88, with higher scores indicating more severe symptoms.
  score on a scale | 171.1 [14 to 2327]
Scleroderma Health Assessment Questionnaire (SHAQ) [Median (Full Range); unit: score on a scale] — SHAQ part 1 (Health Assessment Questionnaire-Disability Index; HAQ-DI) overall score ranges from 0 (without any difficulty) to 3 (unable to do).
  SHAQ part 2 consists of 6 visual analogue scales (VAS) each ranging from 0 (better outcome) to 10 (worse outcome).
  * Pain (SHAQ-VAS-Pain)
  * Intestinal (SHAQ-VAS-GI)
  * Breathing (SHAQ-VAS-Breathing)
  * Raynaud (SHAQ-VAS-Raynaud)
  * Digital ulcers (SHAQ-VAS-DU)
  * Disease Severity (SHAQ-VAS-Disease Severity) Population: Participants with survey data are included in the analysis.
  score on a scale
    HAQ-DI: number analyzed (Participants) | 11
    HAQ-DI | 1.4 [0.1 to 2.6]
    SHAQ-VAS-Pain: number analyzed (Participants) | 11
    SHAQ-VAS-Pain | 1.2 [0.3 to 3]
    SHAQ-VAS-GI: number analyzed (Participants) | 11
    SHAQ-VAS-GI | 0.8 [0 to 3]
    SHAQ-VAS-Breathing: number analyzed (Participants) | 11
    SHAQ-VAS-Breathing | 0.5 [0 to 2.1]
    SHAQ-VAS-Reynaud: number analyzed (Participants) | 11
    SHAQ-VAS-Reynaud | 0.9 [0 to 2.4]
    SHAQ-VAS-DU: number analyzed (Participants) | 11
    SHAQ-VAS-DU | 1.5 [0 to 2.4]
    SHAQ-VAS-Disease Severity: number analyzed (Participants) | 11
    SHAQ-VAS-Disease Severity | 1.4 [0.6 to 2.7]
Cochin Hand Function Scale [Median (Full Range); unit: score on a scale] — Score range 0-90. Higher scores indicates higher disability. Population: Participants with survey data are included in the analysis.
  score on a scale
    number analyzed (Participants) | 11
    (all) | 21 [0 to 72]
Short Form (SF)-36 [Median (Full Range); unit: score on a scale] — Each domain is on a 0-100 scale. The higher the score the less disability. Population: Participants with survey data are included in the analysis.
  score on a scale
    Physical Functioning: number analyzed (Participants) | 11
    Physical Functioning | 32.5 [5 to 90]
    Physical Role Functioning: number analyzed (Participants) | 11
    Physical Role Functioning | 0 [0 to 75]
    Emotional Role Functioning: number analyzed (Participants) | 11
    Emotional Role Functioning | 100 [0 to 100]
    Energy Fatigue: number analyzed (Participants) | 11
    Energy Fatigue | 30 [0 to 65]
    Mental Health: number analyzed (Participants) | 11
    Mental Health | 76 [8 to 84]
    Social Functioning: number analyzed (Participants) | 11
    Social Functioning | 63 [13 to 88]
    Pain: number analyzed (Participants) | 11
    Pain | 45 [0 to 68]
    General Health: number analyzed (Participants) | 11
    General Health | 30 [5 to 75]
    Health Change: number analyzed (Participants) | 11
    Health Change | 25 [0 to 75]
Raynaud Condition Score [Median (Full Range); unit: score on a scale] — Score range: 0-10, where 10 indicates more active Raynaud phenomenon. Population: Participants with survey data are included in the analysis.
  score on a scale
    number analyzed (Participants) | 11
    (all) | 3 [0 to 10]
Patient Global Assessment [Median (Full Range); unit: score on a scale] — Score range: 0 to 10 (higher scores indicate more severe calcinosis). Population: Participants with survey data are included in the analysis.
  score on a scale
    number analyzed (Participants) | 11
    (all) | 4 [1 to 10]
Physician Global Assessment [Median (Full Range); unit: score on a scale] — Score range: 0 to 10 (higher scores indicate more severe calcinosis). Population: Participants with survey data are included in the analysis.
  score on a scale
    number analyzed (Participants) | 11
    (all) | 5 [1 to 10]
Mawdsley Questionnaire [Median (Full Range); unit: score on a scale] — Score range: 0 to 10 (higher scores indicates higher disability from calcinosis). Population: Participants with survey data are included in the analysis.
  score on a scale
    number analyzed (Participants) | 11
    (all) | 4.83 [1.8 to 9.3]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-related Adverse Events Following Treatment With Oral Treprostinil
Description: Number of participants with treatment-related adverse events following treatment with oral treprostinil at 12 months. We defined adverse event as any untoward medical experience occurring to a subject during a clinical trial whether or not it is related to the study drug.
Time Frame: 12 months
Population: Of the 12 patients enrolled in this study, all received at least one dose of study treatment and were evaluated for safety.
Measure: Count of Participants; unit: Participants
Groups:
- Oral Treprostinil: Treprostinil 0.125 mg TID, increased by 0.125 mg TID every 3 to 4 days as tolerated for 12-month period of time.
Arm/Group | Oral Treprostinil
Number analyzed (Participants) | 12
Participants | 11

2. Primary Outcome: Median Rate of Change of Calcinosis in Radiograph Following Treatment With Oral Treprostinil as Assessed by a Novel Radiographic Scoring System
Description: Median rate of change of calcinosis in radiograph following treatment with oral treprostinil as assessed by the Scleroderma Clinical Trial Consortium (SCTC) radiographic scoring system. Historical average SCTC scores in this patient population have ranged from 4.08 to 472.88, with higher scores indicating more severe symptoms.
  The SCTC radiographic score for calcinosis is a validated radiographic scoring system to assess the severity of calcinosis affecting the hands of patients with SSc that accounts for area coverage, density, and anatomic location, higher scores mean worse calcinosis. Physician rates density and percentage of area for 22 regions of each hand, each deferentially weighted in the overall score; individual region values are multiplied my their weight then summed to create an overall score.
Time Frame: Baseline, month 12
Population: Participants who completed the protocol are included in the analysis.
Measure: Median (Full Range); unit: percent change
Arm/Group | Oral Treprostinil
Number analyzed (Participants) | 5
percent change | 22.2 [5.3 to 85.5]

3. Secondary Outcome: Change in Scleroderma Health Assessment Questionnaire (SHAQ)
Description: The Scleroderma Health Assessment Questionnaire (SHAQ) has two parts.
  The first part is a disability index (DI) that consists of the mean of 8 scores from 8 sections (dressing, arising, eating, walking, hygiene, reach, grip, and activities) ranging from 0 (without any difficulty) to 3 (unable to do), with scores summed and divided by 8. The result is the Health Assessment Questionnaire (HAQ)-DI score, which ranges between 0 and 3.
  The second part consists of 6 visual analogue scales (VAS) each ranging from 0 (better outcome) to 10 (worse outcome).
  * Pain (SHAQ-VAS-Pain)
  * Intestinal (SHAQ-VAS-GI)
  * Breathing (SHAQ-VAS-Breathing)
  * Raynaud (SHAQ-VAS-Raynaud)
  * Digital ulcers (SHAQ-VAS-DU)
  * Disease Severity (SHAQ-VAS-Disease Severity)
Time Frame: Baseline, 12 months
Population: Participants with survey data are included in the analysis.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Oral Treprostinil
Number analyzed (Participants) | 11
score on a scale
  HAQ-DI | 0 [-0.08 to 0.1]
  SHAQ-VAS-Pain | -0.03 [-0.1 to 0.13]
  SHAQ-VAS-GI | 0.03 [0 to 0.25]
  SHAQ-VAS-Breathing | 0 [-0.15 to 0.3]
  SHAQ-VAS-Raynaud | 0 [-0.1 to 0.2]
  SHAQ-VAS-DU | 0 [-0.15 to 0.1]
  SHAQ-VAS-Disease Severity | 0 [-0.05 to 0.1]

4. Secondary Outcome: Change in Cochin Hand Functional Scale
Description: Cochin Hand Functional Scale is a 18-question scale, each question ranges from 0 to 5, with a total score range of 0-90. Higher scores indicates higher disability.
Time Frame: Baseline, 12 months
Population: Participants with survey data are included in the analysis.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Oral Treprostinil
Number analyzed (Participants) | 11
score on a scale | -0.17 [-1 to 4.33]

5. Secondary Outcome: Change in Short Form (SF)-36
Description: The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale. The higher the score the less disability.
Time Frame: Baseline, 12 months
Population: Participants with survey data are included in the analysis.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Oral Treprostinil
Number analyzed (Participants) | 11
score on a scale
  Physical Functioning | 0 [-33.3 to 8.3]
  Physical Role Functioning | 0 [0 to 4.17]
  EMotional Role Functioning | 0 [-33.3 to 5.58]
  Energy and fatigue | 0 [-0.83 to 6.67]
  Mental Health | 1 [-1.33 to 6.67]
  Social Functioning | 0 [-8.33 to 6.17]
  Pain | 0 [-4 to 7.67]
  General Health | 0.42 [-1.67 to 3.33]
  Health Change | 2.08 [0 to 8.33]

6. Secondary Outcome: Change in Mawdsley Calcinosis Questionnaire
Description: Mawdsley Calcinosis Questionnaire is an 18-question survey with an overall score of 0-10; each individual question ranges from 0-10, scores are totaled and averaged to and divided by 18 to create the overall score. Higher scores indicate higher disability from calcinosis.
Time Frame: Baseline, 12 months
Population: Participants with survey data are included in the analysis.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Oral Treprostinil
Number analyzed (Participants) | 11
score on a scale | 2 [1 to 2]

7. Secondary Outcome: Change in Raynaud Condition Score
Description: The Raynaud Condition Score is a single question questionnaire, ranges from 0-10, where 10 indicates more active Raynaud phenomenon. Raynaud is an exaggerated vascular response to cold exposure or emotion with at least a 2-phase color change in finger(s) and often toe(s) consisting of pallor, cyanosis, and/or reactive hyperemia: usually one phase is pallor.
Time Frame: Baseline, 12 months
Population: Participants with survey data are included in the analysis.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Oral Treprostinil
Number analyzed (Participants) | 11
score on a scale | 0 [-0.67 to 0.33]

8. Secondary Outcome: Change in Patient Global Assessment of Calcinosis Severity
Description: Patient global assessment of calcinosis severity at 1 year versus baseline. Score range: 0 to 10 (higher scores indicate more severe calcinosis).
Time Frame: Baseline, 12 months
Population: Participants with survey data are included in the analysis.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Oral Treprostinil
Number analyzed (Participants) | 11
score on a scale | 0 [-0.83 to 0.33]

9. Secondary Outcome: Change in Physician Global Assessment of Calcinosis Severity
Description: Physician global assessment of calcinosis severity at 1 year versus baseline. Score range: 0 to 10 (higher scores indicate more severe calcinosis).
Time Frame: Baseline, 12 months
Population: Participants with survey data are included in the analysis.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Oral Treprostinil
Number analyzed (Participants) | 11
score on a scale | -0.08 [-0.33 to 0.33]

10. Secondary Outcome: Baseline Cortical Area Measured by HR-pQCT in SSc Patients With Calcinosis.
Description: Bone cortical area is a bone microarchitecture measurement assessed by High Resolution peripheral Quantitative Computed Tomography (HRpQCT) at the distal tibia. Lower levels of cortical area are associated with more bone fragility.
Time Frame: Baseline visit (average approximately 3 hours for the scan)
Population: Participants with High Resolution peripheral Quantitative Computed Tomography device (HRpQCT) data were included in the analysis.
Measure: Median (Full Range); unit: mm^2
Arm/Group | Oral Treprostinil
Number analyzed (Participants) | 11
mm^2 | 104.8 [81.5 to 129.3]

11. Secondary Outcome: Baseline Cortical Porosity Measured by HR-pQCT in SSc Patients With Calcinosis.
Description: Bone cortical porosity is a bone microarchitecture measurement assessed by High Resolution peripheral Quantitative Computed Tomography (HRpQCT) at the distal tibia. Higher levels of cortical porosity are associated with more bone fragility.
Time Frame: Baseline visit (average approximately 3 hours for the scan)
Population: as for outcome 10
Measure: Median (Full Range); unit: percentage of void space
Arm/Group | Oral Treprostinil
Number analyzed (Participants) | 11
percentage of void space | 0.034 [0.013 to 0.048]

12. Secondary Outcome: Number of Patients With Changes in Vascular and SSc-Pulmonary Arterial Hypertension (PAH) Associated Biomarkers Following Treatment With Treprostinil at 1 Year Compared to Baseline
Description: SSc-PAH associated biomarkers following treatment with treprostinil at 1 year compared to baseline. Ang-1 Ang-2 MMP-2, MMP-9 NT-proBNP, PIGF VEGFR1, sRAGE GLUT-1 Ficolin-1 MBL H62 plex (includes VEGF, PDGFBB, bFGF,IL-13, HGF, IL-6, IL-1β, IL-2, IL-4, IL-5, IL-8, IL-10, IL-12, IL-13,[TNF]-α,[IFN]-γ)
Time Frame: 12 months
Population: Data were not collected for this outcome measure.
Arm/Group | Oral Treprostinil
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected every 3 months up to 12 months and at 13 months from enrollment (3 months, 6 months, 9 month, 12 month and 13 months).
Description: Adverse event and serious adverse event were defined as per clinicaltrials.gov definitions.
Arm/Group | Oral Treprostinil
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 11/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Treprostinil (N=12)
Headache (Nervous system disorders) | 8
Abdominal Pain (Gastrointestinal disorders) | 6
Diarrhea (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 3
Flushing (General disorders) | 2
Jaw Pain (Musculoskeletal and connective tissue disorders) | 2
dizziness (General disorders) | 2
hypotension (Cardiac disorders) | 1 — Defined as systolic blood pressure < 90 or diastolic blood pressure < 60 mmHg
epistaxis (Ear and labyrinth disorders) | 1
weight loss (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-01): https://cdn.clinicaltrials.gov/large-docs/95/NCT02663895/Prot_SAP_000.pdf